CLINICAL TRIAL: NCT01158937
Title: Pharmacokinetic Study of Extended Infusion Meropenem in Adult Cystic Fibrosis Patient With Exacerbation of Pulmonary Infection
Brief Title: Pharmacokinetic Study of Extended Infusion Meropenem in Adult Cystic Fibrosis Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate enrolment and lack of resources
Sponsor: Unity Health Toronto (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: REB#08-316
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Cystic Fibrosis Pulmonary Exacerbation
Keywords: meropenem; cystic fibrosis; extended infusion; pharmacokinetic
MeSH Terms: conditions — Cystic Fibrosis | interventions — Meropenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extended Meropenem Infusion (Experimental): Meropenem Infusion over 3 hours
  Interventions: Drug: Meropenem Infusion
- Bolus Meropenem Infusion (Experimental): Meropenem infusion over 30 minutes
  Interventions: Drug: Meropenem Infusion

INTERVENTIONS:
Drug: Meropenem Infusion — Meropenem 2g infused intravenously over 30 mins (bolus infusion) Meropenem 2g infused intravenously over 3 hours (extended infusion)
  Other Names: Meropenem or Merrem(R)

SUMMARY:
Meropenem is an intravenous antibiotic commonly used to treat acute exacerbation of respiratory infections in cystic fibrosis. The research study aims to determine if a different method of infusing the drug over 3 hours or longer, instead of the traditional half-hour will improve target attainment of drug concentrations and bactericidal activity. A secondary aim is to assess if the pharmacokinetics of meropenem is different during active infection compared to non-infective stage. Twelve patients admitted with acute respiratory infection and who requires meropenem will be enrolled into the study. Meropenem blood concentrations collected over 8 hours will be measured after half-hour and 3-hour infusions on different days. A pharmacokinetic modelling and Monte Carlo simulation program will use the data to assess and predict the optimal method of dosing. When patients return for a follow-up clinic visit, a single dose of meropenem will be administered and blood concentrations will be measured to determine the pharmacokinetics during non-infective stage.

DETAILED DESCRIPTION:
Meropenem plays a crucial role in the treatment of pulmonary exacerbations in cystic fibrosis patients, because it has activity against both P. aeruginosa and B. cepacia, two of the most problematic pathogens that are encountered in this disease. These organisms cause chronic endobronchitis with frequent exacerbations which lead to significant morbidity and premature mortality. Treatment options for pulmonary exacerbations are limited due to the high rates of resistance with currently available antibiotics and lack of development of new effective antibiotics. Therefore optimization of the dosing of meropenem, by use of extended infusion strategy, is one method to allow us to maximize the efficacy of this drug. Meropenem is a beta-lactam type antibiotic with time-dependent bactericidal activity and hence it is suitable for extended infusion dosing. The key rationale for extended infusion of beta-lactam antibiotics is to allow for optimization of pharmacodynamic target attainment of time above the minimal inhibitory concentrations (T>MIC) to maximize bactericidal killing and optimize clinical outcomes. The use of this infusion strategy has been studied in non-cystic fibrosis patients treated primarily with piperacillin-tazobactam or meropenem for P. aeruginosa infections. The application of this strategy in cystic fibrosis patients has not been well studied, and there is no data for the treatment of B. cepacia infections. Also the pharmacokinetic characteristics of meropenem in adult cystic fibrosis patients with pulmonary exacerbation have not been previously studied. It is unclear whether or not the pharmacokinetic profile of meropenem in patients without exacerbation can be accurately extrapolated to those patients with exacerbation. The first phase of this study will, therefore, describe the pharmacokinetic profile of meropenem and the distribution of MICs for P. aeruginosa and B. cepacia in a population of adult cystic fibrosis patients with pulmonary exacerbation. The data will be used to determine an optimal extended infusion dosing strategy specifically for our patients with cystic fibrosis. The second phase of our study will provide additional data on the pharmacokinetics of meropenem in patients without active infection.

Significance of study:

This study will provide new information regarding the pharmacokinetics of meropenem in a population of cystic fibrosis patients with pulmonary exacerbation. This will allow us to apply Monte Carlo simulation to the data set with greater confidence as it directly reflects our own target population. Optimization of meropenem dosing based on pharmacodynamic profile and Monte Carlo simulation lays the groundwork for clinical efficacy studies in the future. Based on results from previous studies, optimization of meropenem dosing has the potential to produce better patient outcomes, reduce drug utilization and cost and reduce rates of resistance. These can be examined in future clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old,
* currently experiencing new or exacerbation of active pulmonary infection as evidenced by increased coughing, sputum production, wheezing, white blood count and/or fever,
* requires meropenem for treatment,
* recent sputum culture positive for P. aeruginosa and/or B. cepacia at a prior visit,
* be able to provide written informed consent.

Exclusion Criteria:

* hypersensitivity and/or intolerance to meropenem,
* history of seizures,
* current use of valproic acid,
* significant psychiatric illness,
* contraindication to insertion of a venous catheter,
* worsening of clinical status requiring admission to intensive care unit (ICU),
* creatinine clearance ≤50 ml/min,
* significant cystic fibrosis-related liver dysfunction characterized by portal hypertension and cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of extended infusion meropenem in Cystic Fibrosis | Two x eight hour pharmacokinetic monitoring periods (carried over 2 days).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cortes, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada